CLINICAL TRIAL: NCT00412152
Title: A Randomised, Double-blind, Parallel-group, Multicentre Study to Demonstrate Improvement in Symptoms of Constipation in Subjects With Non-malignant Pain Taking Oxycodone Equivalent of >20 mg/Day and <50 mg/Day as Oxycodone/Naloxone Prolonged Release Compared to Subjects Taking Oxycodone Prolonged Release Tablets Alone.
Brief Title: Oxycodone-naloxone in Relieving Opioid-related Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN3001; 2005-002398-57 (EudraCT Number)
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Pain
Keywords: A randomised; double blind; parallel group; multicentre study to demonstrate improvement in symptoms of constipation in subjects with non malignant pain; Moderate to severe chronic non-malignant pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxycodone nalaxone prolonged release tablets (OXN)

SUMMARY:
The primary objective of this study is to demonstrate that subjects with moderate to severe non-malignant pain taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets alone.

DETAILED DESCRIPTION:
Patients with a documented history of moderate to severe non-malignant pain that require around the clock opioid therapy will be randomised to an oxycodone or an oxycodone-naloxone treatment arm to assess the safety and efficacy of oxycodone/naloxone prolonged release compared to oxycodone prolonged-release in relieving opioid-related constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at lest 18 years or older with pain.
* Subjects must report constipation caused or aggravated by opioids.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Subjects with evidence of significant structural abnormalities of the gastrointestinal (GI) tract (e.g. bowel obstruction, strictures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate that subjects with moderate to severe non-malignant pain taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets. | 12 weeks with a 6 month open label extension

CONTACTS AND LOCATIONS:
Overall Officials: Karen Simpson, MBChB, Principal Investigator — Seacroft Hospital, Pain Management Services, L Ward, York Road, Leeds

REFERENCES:
- [Derived] Lowenstein O, Leyendecker P, Lux EA, Blagden M, Simpson KH, Hopp M, Bosse B, Reimer K. Efficacy and safety of combined prolonged-release oxycodone and naloxone in the management of moderate/severe chronic non-malignant pain: results of a prospectively designed pooled analysis of two randomised, double-blind clinical trials. BMC Clin Pharmacol. 2010 Sep 29;10:12. doi: 10.1186/1472-6904-10-12. PMID 20920236
- [Derived] Simpson K, Leyendecker P, Hopp M, Muller-Lissner S, Lowenstein O, De Andres J, Troy Ferrarons J, Bosse B, Krain B, Nichols T, Kremers W, Reimer K. Fixed-ratio combination oxycodone/naloxone compared with oxycodone alone for the relief of opioid-induced constipation in moderate-to-severe noncancer pain. Curr Med Res Opin. 2008 Dec;24(12):3503-12. doi: 10.1185/03007990802584454. PMID 19032132
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN3001